CLINICAL TRIAL: NCT02129322
Title: Effect of Adjuvant Therapy by Sorafenib, Oxaliplatin and S-1o Prevent the Tumor Recurrence for Hepatocellular Carcinoma After Liver Transplantation: A Randomized Controlled Study
Brief Title: Effect of Adjuvant Therapy by Sorafenib, Oxaliplatin and S-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: patients not enrolled
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, First affiliated hospital, Zhejiang University, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYYMedOncoLT01
Record Dates: First submitted 2014-04-28; First posted 2014-05-02 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; S 1 (combination); Oxaliplatin

ARMS (2):
- Sorafenib (Active Comparator): Leading 4 cycles: S-1 + Oxaliplatin Q3W + Sorafenib daily Sequential : Sorafenib maintenance
  Interventions: Drug: Sorafenib; Drug: S-1; Drug: Oxaliplatin
- S-1 and Sorafenib (Experimental): Leading 4 cycles: S-1 + Oxaliplatin Q3W + Sorafenib daily Sequential : 4 cycles of S-1 + Sorafenib maintenance
  Interventions: Drug: Sorafenib; Drug: S-1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Sorafenib
Drug: S-1
Drug: Oxaliplatin

SUMMARY:
The study is designed to investigate the effect of adjuvant therapy by Sorafenib, Oxaliplatin and S-1 to prevent the tumor recurrence for hepatocellular carcinoma after liver transplantation

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma after liver transplantation
* Major organ (heart, lung and brain) function was normal

Exclusion Criteria:

* Any active infectious process
* The presence of clinically confirmed extrahepatic metastasis
* Postoperative dysfunction of any organ

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to Recurrence (TTR) | within five years after liver transplantation
  Time to Recurrence

SECONDARY OUTCOMES:
Overall survival (OS) | within the five years after liver transplantation
  Overall survival

OTHER OUTCOMES:
Circulative tumor cell (CTC) level change | within one year after liver transplantation
  Circulative tumor cell

CONTACTS AND LOCATIONS:
Overall Officials: Weijia fang, Principal Investigator — First Affiliated Hospital,Zhejiang University
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, China